CLINICAL TRIAL: NCT01279018
Title: Persistent Pain After Breast Cancer Treatment With Docetaxel
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Kenneth Geving Andersen, MD, Rigshospitalet, Section for Surgical Pathophysiology
Other Study IDs: H-1-2010-028
Record Dates: First submitted 2011-01-14; First posted 2011-01-19 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2010-06

CONDITIONS: Breast Neoplasms; Pain, Postoperative; Neuralgia; Lymphedema
Keywords: Persistent postsurgical pain; breast cancer; postmastectomy pain syndrome; neuropathic pain
MeSH Terms: conditions — Breast Neoplasms; Pain, Postoperative; Neuralgia; Lymphedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients treated with docetaxel: Patients treated according to the DBCG 07 protocol, that have received docetaxel as part of the adjuvant treatment.

SUMMARY:
Breast cancer treatment is for many patients followed by sequelae, such as persistent pain, sensory disturbances, lymphedema and reduced physical function. These undesired consequences of the treatment are a major clinical problem, with persistent pain affecting 25-60%, sensory disturbances 20-80%, lymphedema 2-86% and reduced physical function 13-28% of patients. Development of persistent pain after breast cancer treatment, involves a complex pathophysiology that involves pre-, intra- and postoperative factors. Several risk factors for the development of persistent pain after breast cancer treatment have been identified; young age, psychosocial factors, surgical procedure and radiation therapy. Neurotoxicity is a well know attribute of many chemotherapeutic agents, such as taxanes. The purpose of this nationwide study is to retrospectively examine a cohort of breast cancer patients treated with docetaxel, to clarify if docetaxel may influence the prevalence and intensity of persistent pain and other sequelae.

ELIGIBILITY:
Inclusion Criteria:

* Treated for primary breast cancer in Denmark 2007-2008
* Age between 18-80 years
* No recurrent cancer
* Female

Exclusion Criteria:

* Previous breast surgery same side (including plastic and reconstructive surgery)
* Bilateral breast surgery
* Recurrent cancer or metastatic cancer

Ages: 18 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients treated for breast cancer in Denmark 2007 and 2008
Sampling Method: Non-Probability Sample
Enrollment: 2490 (Actual)
Dates: Start 2010-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Docetaxel as a risk factor for development of persistent pain | Between 2-3 years post surgery

SECONDARY OUTCOMES:
Prevalence of persistent pain, sensory disturbances, lymphedema and functional limitations | Between 2-3 years post surgery